CLINICAL TRIAL: NCT03350971
Title: Influence of Training With Virtual Reality on Myocardial Revascularization: Randomized Clinical Trial
Brief Title: Influence of Virtual Reality on Myocardial Revascularization
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidade Metodista de Piracicaba (Other)
Responsible Party: Principal Investigator, Rodrigo Santiago Barbosa Rocha, Phd, principal investigator, Universidade Metodista de Piracicaba
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2075500
Record Dates: First submitted 2017-11-12; First posted 2017-11-22 (Actual); Last update posted 2018-03-20 (Actual); Status verified 2018-03

CONDITIONS: Myocardial Infarction
Keywords: virtual reality; physical therapy; myocardial revascualrization
MeSH Terms: conditions — Myocardial Infarction

STUDY DESIGN:
Intervention Model Description: Randomized clinical trial
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Virtual reality training (Experimental): Training with ergometer associated with training on wii videogame during 4 days
  Interventions: Other: Virtual reality training
- Control (Active Comparator): chest physical therapy
  Interventions: Other: Control

INTERVENTIONS:
Other: Virtual reality training — training with Wii games, ergometer exercise, ambulation, standing exercises
  Arms: Virtual reality training
Other: Control — chest physical therapy exercises
  Arms: Control

SUMMARY:
Coronary artery disease is a dysfunction characterized by the narrowing of the coronary arteries in due to the accumulation of atheromatous plaques. The surgery of myocardial revascularization is a surgical procedure of choice performed in individuals with to improve symptoms and survival. Cardiovascular surgeries of this size in an extended time of rest after the procedure. Such immobility may have repercussions to the functionality of the individual. Thus, the early mobilization with the use of reality in the Intensive Care Units (ICU) emerges as a potential means of of complications in the postoperative period of cardiac surgery.

DETAILED DESCRIPTION:
The study will be performed at the ICU coronary artery of the Hospital de Clínicas Gaspar Viana de Belém-Pará. 40 volunteers will participate in the study.

preoperative period of myocardial revascularization. The oxidative stress (by the method called Optical Morphology by Oxidative Stress, using capillary blood drops), the modulation autonomic heart rate (with a Polar® model RS800CX) and motor function (through the Medical Research Council scale), before and after the application of protocol for cardiac rehabilitation with ergometer, virtual reality and ambulation. Volunteers will be randomized into a control group who receive the cardiac rehabilitation protocol from the hospital and the Early Mobilization Group, which will receive the cardiac rehabilitation protocol plus virtual reality training using Wii video game from Nintendo.

ELIGIBILITY:
Inclusion Criteria:

* Male patients over 50 years of age to 80 years
* Body Mass Index (BMI) between 20 and 30 BMI kg / m2
* Candidates for elective and conventional myocardial revascularization surgery
* Hemodynamic stability with or without the use of positive inotropes

Exclusion Criteria:

* Patients with previous pulmonary diseases, with ejection fraction below 35% or greater than 54%
* Undergo concomitant surgeries and who underwent surgical reoperation and intraoperative death
* Also excluded are those with motor and neurological deficits, as well as contraindications for performing 6MWT
* orthopedic limitations
* unstable angina, HR> 120 bpm at rest, systolic pressure> 180 mmHg or diastolic> 100 mmHg.

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2017-01-01 (Actual); Primary Completion 2018-02-01 (Actual); Study Completion 2018-02-01 (Actual)

PRIMARY OUTCOMES:
Cardiac autonomic modulation | 7 days
  Avaliation during aplication of protocol (1 week) of heart rate variability on influence of autonomus nervous system on cardiac function

CONTACTS AND LOCATIONS:
Overall Officials: Rodrigo S Rocha, Doctor, Principal Investigator — Universidade do Estado do Pará
Locations (1):
- Hospital de Clínicas Gaspar Viana, Belém, Pará, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Faber AW, Patterson DR, Bremer M. Repeated use of immersive virtual reality therapy to control pain during wound dressing changes in pediatric and adult burn patients. J Burn Care Res. 2013 Sep-Oct;34(5):563-8. doi: 10.1097/BCR.0b013e3182777904. PMID 23970314
- [Result] Sibilla A, Nydahl P, Greco N, Mungo G, Ott N, Unger I, Rezek S, Gemperle S, Needham DM, Kudchadkar SR. Mobilization of Mechanically Ventilated Patients in Switzerland. J Intensive Care Med. 2020 Jan;35(1):55-62. doi: 10.1177/0885066617728486. Epub 2017 Aug 29. PMID 28847238
- [Result] da Costa Torres D, Dos Santos PM, Reis HJ, Paisani DM, Chiavegato LD. Effectiveness of an early mobilization program on functional capacity after coronary artery bypass surgery: A randomized controlled trial protocol. SAGE Open Med. 2016 Dec 14;4:2050312116682256. doi: 10.1177/2050312116682256. eCollection 2016. PMID 28348739